CLINICAL TRIAL: NCT02073279
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Satralizumab (SA237) as Monotherapy in Patients With Neuromyelitis Optica (NMO) and Neuromyelitis Optica Spectrum Disorder (NMOSD)
Brief Title: Efficacy and Safety Study of Satralizumab (SA237) as Monotherapy to Treat Participants With Neuromyelitis Optica (NMO) and Neuromyelitis Optica Spectrum Disorder (NMOSD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BN40900; SA-309JG (Other: Chugai Pharmaceutical); 2015-005431-41 (EudraCT Number)
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Results first posted 2020-12-31 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-01

CONDITIONS: Neuromyelitis Optica (NMO); NMO Spectrum Disorder (NMOSD)
MeSH Terms: conditions — Neuromyelitis Optica | interventions — satralizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Satralizumab (Experimental): Participants randomized to this arm for the double-blind period will receive satralizumab monotherapy. The double-blind period for the participant ends either when the participant experiences a Clinical Endpoint Committee (CEC) confirmed protocol-defined relapse, the total number of CEC confirmed protocol-defined relapses reaches 44, or 1.5 years after the last patient was randomized. In the open-label extension period, the participant will receive satralizumab SC injection at Weeks 0, 2, and 4, and Q4W thereafter, up to the end of the study.
  Interventions: Drug: Satralizumab
- Placebo (Placebo Comparator): Participants randomized to this arm for the double-blind period will receive placebo monotherapy. The double-blind period for the participant ends either when the participant experiences a Clinical Endpoint Committee (CEC) confirmed protocol-defined relapse, the total number of CEC confirmed protocol-defined relapses reaches 44, or 1.5 years after the last patient was randomized.. In the open-label extension period, the participant will receive satralizumab SC injection at Weeks 0, 2, and 4, and Q4W thereafter, up to the end of the study.
  Interventions: Drug: Satralizumab; Drug: Placebo

INTERVENTIONS:
Drug: Satralizumab — Satralizumab will be administered subcutaneously (SC) at Weeks 0, 2, and 4, and thereafter once every 4 weeks (Q4W).
  Other Names: SA237; RG6168
Drug: Placebo — Placebo will be administered subcutaneously (SC) at Weeks 0, 2, and 4, and thereafter once every 4 weeks (Q4W).
  Arms: Placebo

SUMMARY:
The objectives of this study are to evaluate the efficacy, safety, pharmacodynamic, pharmacokinetic and immunogenic profiles of satralizumab in participants with NMO and NMOSD.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be diagnosed as having either neuromyelitis optica (NMO) or NMO spectrum disorder (NMOSD), defined as the following:

   1. NMO as defined by Wingerchuk et al. 2006 criteria (requires all of the following 3 criteria: I. Optic neuritis, II. Acute myelitis, III. At least two of three supportive criteria: Contiguous spinal cord lesion identified on a magnetic resonance imaging [MRI] scan extending over 3 vertebral segments; Brain MRI not meeting diagnostic criteria for multiple sclerosis [MS]; NMO-IgG seropositive status)
   2. NMOSD as defined by either of following criteria with anti-aquaporin-4 (AQP4) antibody seropositive status at screening: i. Idiopathic single or recurrent events of longitudinally extensive myelitis (≥3 vertebral segment spinal cord MRI lesion); ii. Optic neuritis, single, recurrent or simultaneous bilateral
2. Clinical evidence of at least 1 documented relapse (including first attack) in last 12 months prior to screening
3. Expanded Disability Status Scale (EDSS) score from 0 to 6.5 inclusive at screening
4. Age 18 to 74 years, inclusive at the time of informed consent
5. Ability and willingness to provide written informed consent and to comply with the requirements of the protocol

Exclusion Criteria:

1. Clinical relapse onset (including first attack) within 30 days prior to baseline

   Exclusion Criteria Related to Previous or Concomitant Therapy:
2. Any previous treatment with interleukin 6 (IL-6) inhibitory therapy (e.g., tocilizumab), alemtuzumab, total body irradiation or bone marrow transplantation at any time
3. Any previous treatment with anti-CD20, eculizumab, anti-BLyS monoclonal antibody (e.g., belimumab), any other treatment for prevention of multiple sclerosis (MS) relapse (e.g., interferon, natalizumab, glatiramer acetate, fingolimod, teriflunomide or dimethyl fumarate) within 6 months prior to baseline
4. Any previous treatment with anti-CD4, cladribine, cyclophosphamide or mitoxantrone within 2 years prior to baseline
5. Treatment with any investigational agent within 3 months prior to baseline

   Exclusions for General Safety:
6. Pregnancy or lactation.
7. For participants of reproductive potential, a positive result from a serum pregnancy test at screening, or not willing to use reliable means of contraception (physical barrier [participants or partner] in conjunction with a spermicidal product, contraceptive pill, patch, injectables, intrauterine device or intrauterine system) during the treatment period and for at least 3 months after the last dose of study drug
8. Any surgical procedure (except for minor surgeries) within 4 weeks prior to baseline
9. Evidence of other demyelinating disease or progressive multifocal leukoencephalopathy (PML)
10. Evidence of serious uncontrolled concomitant diseases that may preclude participant participation, as described; Other nervous system disease, cardiovascular disease, hematologic/hematopoiesis disease, respiratory disease, muscular disease, endocrine disease, renal/urologic disease, digestive system disease, congenital or acquired severe immunodeficiency
11. Known active infection (excluding fungal infections of nail beds or caries dentium) within 4 weeks prior to baseline
12. Evidence of chronic active hepatitis B or C
13. History of drug or alcohol abuse within 1 year prior to baseline
14. History of diverticulitis that, in the Investigator's opinion, may lead to increased risk of complications such as lower gastrointestinal perforation
15. Evidence of active tuberculosis (excluding participants receiving chemoprophylaxis for latent tuberculosis infection)
16. Evidence of active interstitial lung disease
17. Receipt of any live or live attenuated vaccine within 6 weeks prior to baseline
18. History of malignancy within the last 5 years, including solid tumors, hematologic malignancies and in situ carcinoma (except basal cell and squamous cell carcinomas of the skin, or in situ carcinoma of the cervix uteri that have been completely excised and cured)
19. History of severe allergic reaction to a biologic agent (e.g., shock, anaphylactic reactions)
20. Active suicidal ideation within 6 months prior to screening, or history of suicide attempt within 3 years prior to screening
21. History of Stevens-Johnson syndrome
22. Following laboratory abnormalities at screening*.

    1. White blood cells <3.0 x10^3/microliter (μL)
    2. Absolute neutrophil count <2.0 x 10^3 /μL
    3. Absolute lymphocyte count <0.5 x 10^3 /μL
    4. Platelet count <10 x 10^4 /μL
    5. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 times the upper limit of normal.

       * If retest is conducted, the last value of retest before randomization must meet study criteria.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2014-08-05 (Actual); Primary Completion 2018-10-12 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (58):
- United States (20):
  - University of Colorado Denver -; Neurology, Aurora, Colorado
  - University of Miami UHealth Professional Arts Center, Miami, Florida
  - The MS Center of Vero Beach, Vero Beach, Florida
  - Columbus Research and Wellness, Columbus, Georgia
  - University of Chicago; Neurology, Chicago, Illinois
  - Consultants in Neurology Ltd, Northbrook, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - MidAmerica Neuroscience Institute, Prairie Village, Kansas
  - University of Michigan Health System, Ann Arbor, Michigan
  - Wayne State University - Comp Clinic and MS. Center, Detroit, Michigan
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Neurological Institute PA, Charlotte, North Carolina
  - OhioHealth Research Institute, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - UT Medicine San Antonio, San Antonio, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - Wheaton Franciscan Healthcare - St. Francis Outpatient Center; Center for Neurological Disorders, Milwaukee, Wisconsin
- Bulgaria (5):
  - Medical Help Center EOOD, Dobrich
  - MMA-MHAT Pleven - Clinic for Neurology, Pleven
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - MHATNP Sveti Naum EAD, Sofia
  - UMHAT Alexandrovska, EAD, Sofia
- Canada (3):
  - MS Clinical Trials Group, Vancouver, British Columbia
  - Recherche Sepmus Inc., Greenfield Park, Quebec
  - Centre hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
- Klinicki bolnicki centar Osijek, Osijek, Croatia
- Georgia (3):
  - LTD Helsicore, Tbilisi
  - Pineo Medical Ecosystem LTD, Tbilisi
  - S.Khechinashvili Tbilisi State Medical University Clinic Ne, Tbilisi
- PO G.Rodolico, AOU Policlinico-Vittorio Emanuele Catania, Catania, Sicily, Italy
- Malaysia (2):
  - Hospital Universiti Sains Malaysia [Neurology], Kubang Kerian, Kelantan
  - Hospital Kuala Lumpur, Kuala Lumpur
- Philippine General Hospital, Manila, Philippines
- Poland (2):
  - NZOZ Wielospecjalistyczna Poradnia Lekarska SYNAPSIS, Katowice
  - Miedzyleski Szpital Specjalistyczny w Warszawie, Warsaw
- San Juan MS Center, Guaynabo, Puerto Rico
- SC Clubul Sanatatii SRL, Campulung Muscel, Romania
- South Korea (4):
  - Korea University Anam Hospital - Neurology, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Severance Hospital - Yonsei University Health System - Neurology, Seoul
- Taiwan (3):
  - China Medical University Healthcare System, Taichung
  - National Cheng Kung University Hospital; Neurology, Tainan
  - Taipei Veterans General Hospital-Neurology, Taipei
- Turkey (Türkiye) (2):
  - Bilim University Medical Faculty Florence Nightingale Hospital, Istanbul
  - Ondokuz Mayis Univ. Med. Fac., Samsun
- Ukraine (9):
  - Ivano-Frankivska oblasna klinichna likarnia, Ivano-Frankivsk, KIEV Governorate
  - Ivano-Frankivska miska klinichna likarnia №1, Ivano-Frankivsk, KIEV Governorate
  - Kiev National Medical University, Kiev, KIEV Governorate
  - Municipal Foundation of Kyiv Regional Council " Kyiv Region, Kyiv, KIEV Governorate
  - Reginal clinical psyconeurological hospital, Ternopil, KIEV Governorate
  - Vinnytskyi natsionalnyi medychnyi universytet imeni M.I. Pyr, Vinnytsia, Poltava Governorate
  - Municipal Establishment "City Clinical Hospital #2; Neurology, Zaporozhya, Poltava Governorate
  - Miska Klinichna Likarnia №16, Dnipropetrovsk, Tavria Okruha
  - KU "Odeskyi oblasnyi medychnyi tsentr psykhichnoho zdorovia", Odesa, Tavria Okruha

REFERENCES:
- [Derived] Bennett JL, Fujihara K, Saiz A, Traboulsee AL, Greenberg BM, Weinshenker BG, Patti F, Kleiter I, Palace J, De Seze J, Evans R, Blondeau K, Klingelschmitt G, Vodopivec I, Rahim M, Yamamura T. Long-Term Efficacy and Safety of Satralizumab in Patients With Neuromyelitis Optica Spectrum Disorder From the SAkuraMoon Open-Label Extension Study. Neurol Neuroimmunol Neuroinflamm. 2025 Sep;12(5):e200450. doi: 10.1212/NXI.0000000000200450. Epub 2025 Jul 31. PMID 40743487
- [Derived] Greenberg BM, Fujihara K, Weinshenker B, Patti F, Kleiter I, Bennett JL, Palace J, Blondeau K, Burdeska A, Ngwa I, Klingelschmitt G, Triyatni M, Yamamura T. Analysis of infection rates in neuromyelitis optica spectrum disorder: Comparing satralizumab treatment in SAkuraMoon, post-marketing, and US-based health claims data. Mult Scler Relat Disord. 2025 Jul;99:106444. doi: 10.1016/j.msard.2025.106444. Epub 2025 Apr 19. PMID 40288333
- [Derived] Kleiter I, Traboulsee A, Palace J, Yamamura T, Fujihara K, Saiz A, Javed A, Mayes D, Budingen HV, Klingelschmitt G, Stokmaier D, Bennett JL. Long-term Efficacy of Satralizumab in AQP4-IgG-Seropositive Neuromyelitis Optica Spectrum Disorder From SAkuraSky and SAkuraStar. Neurol Neuroimmunol Neuroinflamm. 2022 Dec 8;10(1):e200071. doi: 10.1212/NXI.0000000000200071. Print 2023 Jan. PMID 36724181
- [Derived] Yamamura T, Weinshenker B, Yeaman MR, De Seze J, Patti F, Lobo P, von Budingen HC, Kou X, Weber K, Greenberg B. Long-term safety of satralizumab in neuromyelitis optica spectrum disorder (NMOSD) from SAkuraSky and SAkuraStar. Mult Scler Relat Disord. 2022 Oct;66:104025. doi: 10.1016/j.msard.2022.104025. Epub 2022 Jul 5. PMID 36007339
- [Derived] Traboulsee A, Greenberg BM, Bennett JL, Szczechowski L, Fox E, Shkrobot S, Yamamura T, Terada Y, Kawata Y, Wright P, Gianella-Borradori A, Garren H, Weinshenker BG. Safety and efficacy of satralizumab monotherapy in neuromyelitis optica spectrum disorder: a randomised, double-blind, multicentre, placebo-controlled phase 3 trial. Lancet Neurol. 2020 May;19(5):402-412. doi: 10.1016/S1474-4422(20)30078-8. PMID 32333898

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Double-blind (DB) period lasted up to the primary clinical cut-off date (CCOD: 12 Oct 2018) when the study reached 1.5 years since the date of randomization of the last participant enrolled.
  The Open Label Period lasted up to clinical cut-off date (31-Jan-2022).
Pre-assignment Details: Participants with neuromyelitis optica (NMO) or NMO spectrum disorder (NMOSD) were randomized 2:1 to receive either satralizumab 120 mg or matching placebo.
Groups:
- Placebo, Then Satralizumab: Participants received matching placebo, subcutaneous (SC) injection at Weeks 0, 2 and 4, and every 4 weeks (Q4W) thereafter throughout the double-blind (DB) period up to protocol-defined relapse. Following the DB period, all participants received satralizumab 120 mg SC injection at Weeks 0, 2 and 4, and Q4W thereafter up to the clinical cut-off date (CCOD). At the CCOD, participants who had not experienced a relapse during the DB period were invited to initiate satralizumab 120 mg SC injection (at Weeks 0, 2 and 4, and Q4W thereafter) after 4 weeks from their last study treatment dose in the DB period.
- Satralizumab, Then Satralizumab: Participants received satralizumab 120 mg subcutaneous (SC) injection at Weeks 0, 2 and 4, and every 4 weeks (Q4W) thereafter throughout the double-blind (DB) period. Participants who experienced a protocol defined relapse could continue in the Open Label Extension (OLE) period 31 days after relapse. Participants who completed the DB period without relapse could participate in the OLE period 4 weeks after receiving their last dose in the DB period. All OLE participants received satralizumab 120 mg SC injection at Weeks 0, 2 and 4, and Q4W thereafter.
Period: Double-blind Period
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Started | 32 | 63
Completed (Double-blind Period) | 28 | 56
Not Completed | 4 | 7
Not completed — Adverse Event | 1 | 1
Not completed — Switched to another treatment | 1 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Refused Treatment/Did Not Cooperate | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2
Period: Open-label Extension Period
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Started | 28 | 56
Completed | 21 | 41
Not Completed | 7 | 15
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 0 | 4
Not completed — Switched to another treatment | 1 | 4
Not completed — Protocol Violation | 0 | 1
Not completed — Refused Treatment/Did Not Cooperate | 0 | 1
Not completed — Withdrawal by Subject | 4 | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants randomized to the treatment groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab | Total
Number analyzed (Participants) | 32 | 63 | 95
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.5 (10.5) | 45.3 (12.0) | 43.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 46 | 77
  Male | 1 | 17 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 9 | 12
  Not Hispanic or Latino | 28 | 50 | 78
  Not Stated | 0 | 4 | 4
  Unknown | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 6 | 8 | 14
  Black or African American | 3 | 13 | 16
  White | 22 | 37 | 59
  Other | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to First Protocol-Defined Relapse (TFR) During the Double-Blind (DB) Period
Description: TFR was defined as time from randomization to first occurrence of relapse in the DB period. Protocol-defined relapse was occurrence of new or worsening neurological symptoms attributable to neurological neuromyelitis optica (NMO) or neuromyelitis optica spectrum disorder (NMOSD). Symptoms had to persist for >24 hours and not be attributable to confounding clinical factors (e.g., fever, infection, injury, change in mood, adverse reactions to medications). New or worsening neurological symptoms that occurred < 31 days following onset of a protocol-defined relapse were considered part of same relapse (i.e., if 2 relapses had onset days that were 30 days of one another, they were counted only as 1 relapse), and onset date used in analysis was the date of first relapse.
Time Frame: Up to Week 216
Population: ITT population included all participants randomized to the treatment groups. For participants who had not relapsed, the TFR was censored on the date of end of the DB period.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 63
weeks | 128.3 [29.9 to NA] — Upper limit of CI was not reached due to low number of participants with events. | NA [135.7 to NA] — Median was not reached due to low number of participants with events. Upper limit of CI was not reached due to low number of participants with events.
Statistical Analysis 1: Comparison: Placebo, Then Satralizumab vs Satralizumab, Then Satralizumab; Stratified by prior therapy (B-cell depleting therapy or immunosuppressants/others) and most recent attack (first attack or relapse); Test type: Superiority; p = 0.0184, Log Rank; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.23 to 0.89]

2. Secondary Outcome: Change From Baseline to Week 24 in Visual Analogue Scale (VAS) for Pain During the DB Period
Description: The VAS is a subjective measure of pain consisting of a 100 mm line with two endpoints representing 0 = "no pain" and 100 = "pain as bad as it could be". Participants rated their pain by placing a mark on the line corresponding to their current level of pain. The distance along the line from the "no pain" marker was measured with a ruler giving a pain score out of 100. A higher score indicated more pain and lower scores reflected a better health state. A negative change from baseline indicates an improvement. ANCOVA was used for analysis to report the adjusted mean and standard error (SE).
Time Frame: Baseline, Week 24
Population: ITT population included all participants randomized to the treatment groups. Number analyzed is the number of participants with data available for analyses at the given timepoint. Missing data were imputed by BOCF method.
Measure: Mean (Standard Error); unit: score on scale
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 62
score on scale
  Baseline | 27.563 (5.438) | 31.661 (3.665)
  Change from Baseline to Week 24 | -5.949 (4.832) | -2.735 (4.260)
Statistical Analysis 1: Comparison: Placebo, Then Satralizumab vs Satralizumab, Then Satralizumab; Test type: Superiority; p = 0.4436, ANCOVA; ANCOVA model: treatment group as fixed effect and baseline measurements, prior therapy, most recent attack (first attack/relapse) as covariates; Mean Difference (Final Values) = 3.215, 95% CI [-5.086 to 11.515], Standard Error of Mean 4.178

3. Secondary Outcome: Change From Baseline to Week 24 in Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale During the DB Period
Description: The FACIT Fatigue scale is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function over the past 7 days. As each of the 13 items of the scale ranges from 0-4, the range of possible scores was computed using FACIT scoring algorithm as 0-52, where 0 is the worst possible score and 52 the best which indicated less fatigue. A positive change from baseline indicates an improvement.
Time Frame: Baseline, Week 24
Population: ITT population included all participants randomized to the treatment groups. Number analyzed is the number of participants with data available for analyses at the given timepoint. Missing data was imputed using BOCF method
Measure: Mean (Standard Error); unit: score on scale
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 62
score on scale
  Baseline | 29.656 (2.280) | 30.590 (1.492)
  Change from Baseline to Week 24 | 3.602 (1.820) | 5.709 (1.610)
Statistical Analysis 1: Comparison: Placebo, Then Satralizumab vs Satralizumab, Then Satralizumab; Test type: Superiority; p = 0.1824, ANCOVA; ANCOVA model included treatment group as fixed effect. Baseline measurements, prior therapy, most recent attack (first attack/relapse) as covariates; Mean Difference (Final Values) = 2.107, 95% CI [-1.008 to 5.221], Standard Error of Mean 1.567

4. Secondary Outcome: Relapse-Free Rate During the DB Period
Description: Protocol-defined relapse was occurrence of new or worsening neurological symptoms attributable to neurological neuromyelitis optica (NMO) or neuromyelitis optica spectrum disorder (NMOSD). Symptoms had to persist for >24 hours and not be attributable to confounding clinical factors (e.g., fever, infection, injury, change in mood, adverse reactions to medications). New or worsening neurological symptoms that occurred < 31 days following onset of a protocol-defined relapse were considered part of same relapse (i.e., if 2 relapses had onsets within 30 days of one another, they were counted as 1), and onset date used in analysis was the date of first relapse.
Time Frame: Up to Week 216
Population: ITT population included all participants randomized to the treatment groups.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 23 | 56
percentage of participants
  Week 12 | 74.87 | 88.89
  Week 24 | 71.61 | 85.71
  Week 36 | 61.85 | 79.37
  Week 48 | 61.85 | 76.13
  Week 72 | 51.21 | 74.40
  Week 96 | 51.21 | 72.14
  Week 120 | 51.21 | 72.14
  Week 144 | 34.14 | 62.80
  Week 168 | 34.14 | 62.80
  Week 192 | 34.14 | 62.80
  Week 216: number analyzed (Participants) | 23 | 0
  Week 216 | 34.14 |

5. Secondary Outcome: Annualized Relapse Rate (ARR) During the DB Period
Description: The ARR is calculated as the total number of participants with adjudicated PDRs experienced divided by the patient-years at risk. Protocol-defined relapse was occurrence of new or worsening neurological symptoms attributable to neurological NMO or NMOSD. Symptoms had to persist for >24 hours and not be attributable to confounding clinical factors (e.g., fever, infection, injury, change in mood, adverse reactions to medications). New or worsening neurological symptoms that occurred < 31 days following onset of a protocol-defined relapse were considered part of same relapse (2 relapses with onset days in 30 days of one another was counted as 1 relapse), onset date used in analysis was the date of first relapse.
Time Frame: Up to Week 216
Population: ITT population included all participants randomized to the treatment groups.
Measure: Number (95% Confidence Interval); unit: patients w PDRs/patient-years at risk
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 63
patients w PDRs/patient-years at risk | 0.41 [0.24 to 0.67] | 0.17 [0.10 to 0.26]

6. Secondary Outcome: Change From Baseline in Short Form Generic Health Survey (SF-36) Bodily Pain Domain Scores at 24 Week Intervals During the DB Period
Description: The SF-36v2 is a multi-purpose, short form health survey with 36 questions. It has 8 domains (vitality, physical functioning, bodily pain, general health, role-physical, role emotional, social role functioning and mental health) of functional health and well-being scores as well as psychometrically based physical and mental health component summary measures and a preference-based health utility index. The domain scores were transformed to a 0-100 scale, where higher scores indicate better quality of life. A positive change from baseline indicates an improvement.
Time Frame: Baseline up to Week 216
Population: ITT population included all participants randomized to the treatment groups. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 62
score on scale
  Baseline | 42.86 (11.28) | 43.20 (11.08)
  Change from Baseline at Week 24: number analyzed (Participants) | 20 | 54
  Change from Baseline at Week 24 | -0.89 (8.35) | -0.13 (8.09)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 46
  Change from Baseline at Week 48 | 1.75 (5.42) | 1.36 (8.89)
  Change from Baseline at Week 72: number analyzed (Participants) | 13 | 43
  Change from Baseline at Week 72 | 3.19 (8.04) | 0.91 (9.23)
  Change from Baseline at Week 96: number analyzed (Participants) | 8 | 31
  Change from Baseline at Week 96 | 3.43 (5.60) | 2.38 (7.82)
  Change from Baseline at Week 120: number analyzed (Participants) | 3 | 16
  Change from Baseline at Week 120 | 0.00 (8.07) | 0.53 (6.21)
  Change from Baseline at Week 144: number analyzed (Participants) | 2 | 12
  Change from Baseline at Week 144 | -2.22 (8.84) | 2.59 (6.66)
  Change from Baseline at Week 168: number analyzed (Participants) | 1 | 10
  Change from Baseline at Week 168 | 0.80 (NA) — Standard Deviation (SD) was not calculable for 1 participant. | 4.19 (7.01)
  Change from Baseline at Week 192: number analyzed (Participants) | 1 | 2
  Change from Baseline at Week 192 | -8.47 (NA) — SD was not calculable for 1 participant. | 0 (0)
  Change from Baseline at Week 216: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 216 | -12.50 (NA) — SD was not calculable for 1 participant. |

7. Secondary Outcome: Change From Baseline in SF-36 General Health Domain Scores at 24 Week Intervals During the DB Period
Description: as for outcome 6
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 62
score on scale
  Baseline | 39.43 (9.50) | 39.72 (10.41)
  Change from Baseline at Week 24: number analyzed (Participants) | 20 | 54
  Change from Baseline at Week 24 | -0.52 (9.96) | 0.49 (6.46)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 46
  Change from Baseline at Week 48 | 1.85 (9.72) | 1.01 (7.61)
  Change from Baseline at Week 72: number analyzed (Participants) | 13 | 43
  Change from Baseline at Week 72 | 4.83 (12.41) | 3.21 (6.57)
  Change from Baseline at Week 96: number analyzed (Participants) | 8 | 31
  Change from Baseline at Week 96 | 6.60 (9.10) | 3.45 (6.42)
  Change from Baseline at Week 120: number analyzed (Participants) | 3 | 16
  Change from Baseline at Week 120 | 8.72 (13.55) | 3.60 (7.02)
  Change from Baseline at Week 144: number analyzed (Participants) | 2 | 12
  Change from Baseline at Week 144 | 5.23 (14.11) | 2.82 (8.00)
  Change from Baseline at Week 168: number analyzed (Participants) | 1 | 10
  Change from Baseline at Week 168 | -7.13 (NA) — SD was not calculable for 1 participant. | 5.04 (9.45)
  Change from Baseline at Week 192: number analyzed (Participants) | 1 | 2
  Change from Baseline at Week 192 | -4.75 (NA) — SD was not calculable for 1 participant. | 8.32 (11.77)
  Change from Baseline at Week 216: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 216 | -4.75 (NA) — SD was not calculable for 1 participant. |

8. Secondary Outcome: Change From Baseline in SF-36 Mental Health Domain Scores at 24 Week Intervals During the DB Period
Description: as for outcome 6
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 62
score on scale
  Baseline | 42.86 (12.69) | 46.78 (10.10)
  Change from Baseline at Week 24: number analyzed (Participants) | 20 | 54
  Change from Baseline at Week 24 | 0.79 (9.02) | 1.84 (7.05)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 46
  Change from Baseline at Week 48 | -0.58 (7.32) | 2.67 (7.89)
  Change from Baseline at Week 72: number analyzed (Participants) | 13 | 43
  Change from Baseline at Week 72 | 2.62 (6.32) | 1.95 (7.85)
  Change from Baseline at Week 96: number analyzed (Participants) | 8 | 31
  Change from Baseline at Week 96 | -3.60 (6.08) | 2.36 (7.38)
  Change from Baseline at Week 120: number analyzed (Participants) | 3 | 16
  Change from Baseline at Week 120 | -2.62 (6.92) | 0.82 (10.32)
  Change from Baseline at Week 144: number analyzed (Participants) | 2 | 12
  Change from Baseline at Week 144 | 1.31 (1.85) | 2.83 (9.43)
  Change from Baseline at Week 168: number analyzed (Participants) | 1 | 10
  Change from Baseline at Week 168 | 5.23 (NA) — SD was not calculable for 1 participant. | 2.62 (8.89)
  Change from Baseline at Week 192: number analyzed (Participants) | 1 | 2
  Change from Baseline at Week 192 | -13.08 (NA) — SD was not calculable for 1 participant. | -3.93 (12.95)
  Change from Baseline at Week 216: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 216 | -2.62 (NA) — SD was not calculable for 1 participant. |

9. Secondary Outcome: Change From Baseline in SF-36 Physical Functioning Domain Scores at 24 Week Intervals During the DB Period
Description: as for outcome 6
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 62
score on scale
  Baseline | 38.70 (12.24) | 39.48 (10.99)
  Change from Baseline at Week 24: number analyzed (Participants) | 20 | 54
  Change from Baseline at Week 24 | 2.20 (4.62) | 1.96 (6.12)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 46
  Change from Baseline at Week 48 | 2.34 (6.90) | 3.33 (6.76)
  Change from Baseline at Week 72: number analyzed (Participants) | 13 | 43
  Change from Baseline at Week 72 | 6.62 (9.71) | 2.99 (6.94)
  Change from Baseline at Week 96: number analyzed (Participants) | 8 | 31
  Change from Baseline at Week 96 | 5.50 (9.62) | 3.59 (7.49)
  Change from Baseline at Week 120: number analyzed (Participants) | 3 | 16
  Change from Baseline at Week 120 | 7.01 (8.63) | 1.94 (8.05)
  Change from Baseline at Week 144: number analyzed (Participants) | 2 | 12
  Change from Baseline at Week 144 | 4.79 (9.48) | 3.19 (10.87)
  Change from Baseline at Week 168: number analyzed (Participants) | 1 | 10
  Change from Baseline at Week 168 | 1.91 (NA) — SD was not calculable for 1 participant. | -0.96 (8.62)
  Change from Baseline at Week 192: number analyzed (Participants) | 1 | 2
  Change from Baseline at Week 192 | -1.92 (NA) — SD was not calculable for 1 participant. | 4.78 (4.06)
  Change from Baseline at Week 216: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 216 | -3.83 (NA) — SD was not calculable for 1 participant. |

10. Secondary Outcome: Change From Baseline in SF-36 Role-Emotional Domain Scores at 24 Week Intervals During the DB Period
Description: as for outcome 6
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 62
score on scale
  Baseline | 42.24 (13.09) | 42.07 (13.62)
  Change from Baseline at Week 24: number analyzed (Participants) | 20 | 54
  Change from Baseline at Week 24 | -1.57 (15.67) | 3.87 (11.27)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 46
  Change from Baseline at Week 48 | 0.78 (8.57) | 2.73 (10.30)
  Change from Baseline at Week 72: number analyzed (Participants) | 13 | 43
  Change from Baseline at Week 72 | 4.55 (7.96) | 3.89 (9.22)
  Change from Baseline at Week 96: number analyzed (Participants) | 8 | 31
  Change from Baseline at Week 96 | 3.05 (11.98) | 1.12 (11.87)
  Change from Baseline at Week 120: number analyzed (Participants) | 3 | 16
  Change from Baseline at Week 120 | -12.77 (14.07) | 1.31 (14.04)
  Change from Baseline at Week 144: number analyzed (Participants) | 2 | 12
  Change from Baseline at Week 144 | -12.19 (17.23) | 1.74 (13.40)
  Change from Baseline at Week 168: number analyzed (Participants) | 1 | 10
  Change from Baseline at Week 168 | 0.00 (NA) — SD was not calculable for 1 participant. | -0.35 (11.89)
  Change from Baseline at Week 192: number analyzed (Participants) | 1 | 2
  Change from Baseline at Week 192 | -13.93 (NA) — SD was not calculable for 1 participant. | -3.49 (4.93)
  Change from Baseline at Week 216: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 216 | -10.45 (NA) — SD was not calculable for 1 participant. |

11. Secondary Outcome: Change From Baseline in SF-36 Role-Physical Domain Scores at 24 Week Intervals During the DB Period
Description: as for outcome 6
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 62
score on scale
  Baseline | 37.86 (11.28) | 37.43 (11.55)
  Change from Baseline at Week 24: number analyzed (Participants) | 20 | 54
  Change from Baseline at Week 24 | 3.14 (9.92) | 3.52 (8.38)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 46
  Change from Baseline at Week 48 | 4.12 (7.24) | 5.01 (8.25)
  Change from Baseline at Week 72: number analyzed (Participants) | 13 | 43
  Change from Baseline at Week 72 | 5.70 (7.65) | 4.59 (8.56)
  Change from Baseline at Week 96: number analyzed (Participants) | 8 | 31
  Change from Baseline at Week 96 | 5.62 (6.35) | 4.83 (8.31)
  Change from Baseline at Week 120: number analyzed (Participants) | 3 | 16
  Change from Baseline at Week 120 | 2.25 (8.99) | 3.18 (9.46)
  Change from Baseline at Week 144: number analyzed (Participants) | 2 | 12
  Change from Baseline at Week 144 | -3.37 (11.12) | 2.43 (8.80)
  Change from Baseline at Week 168: number analyzed (Participants) | 1 | 10
  Change from Baseline at Week 168 | 0.00 (NA) — SD was not calculable for 1 participant. | 0.00 (9.10)
  Change from Baseline at Week 192: number analyzed (Participants) | 1 | 2
  Change from Baseline at Week 192 | -6.74 (NA) — SD was not calculable for 1 participant. | 4.49 (6.35)
  Change from Baseline at Week 216: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 216 | -17.97 (NA) — SD was not calculable for 1 participant. |

12. Secondary Outcome: Change From Baseline in SF-36 Social Role Functioning Domain Scores at 24 Week Intervals During the DB Period
Description: as for outcome 6
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 62
score on scale
  Baseline | 42.93 (13.22) | 41.01 (11.66)
  Change from Baseline at Week 24: number analyzed (Participants) | 20 | 54
  Change from Baseline at Week 24 | 1.76 (12.42) | 2.42 (9.63)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 46
  Change from Baseline at Week 48 | 0.56 (10.59) | 2.62 (8.17)
  Change from Baseline at Week 72: number analyzed (Participants) | 13 | 43
  Change from Baseline at Week 72 | 0.39 (11.66) | 3.96 (7.93)
  Change from Baseline at Week 96: number analyzed (Participants) | 8 | 31
  Change from Baseline at Week 96 | 0.63 (1.77) | 3.56 (7.89)
  Change from Baseline at Week 120: number analyzed (Participants) | 3 | 16
  Change from Baseline at Week 120 | -5.01 (13.26) | 0.31 (8.48)
  Change from Baseline at Week 144: number analyzed (Participants) | 2 | 12
  Change from Baseline at Week 144 | 7.52 (10.63) | 3.76 (14.68)
  Change from Baseline at Week 168: number analyzed (Participants) | 1 | 10
  Change from Baseline at Week 168 | -5.01 (NA) — SD was not calculable for 1 participant. | -1.50 (7.86)
  Change from Baseline at Week 192: number analyzed (Participants) | 1 | 2
  Change from Baseline at Week 192 | -5.01 (NA) — SD was not calculable for 1 participant. | -2.51 (3.54)
  Change from Baseline at Week 216: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 216 | 0.00 (NA) — SD was not calculable for 1 participant. |

13. Secondary Outcome: Change From Baseline in SF-36 Vitality Domain Scores at 24 Week Intervals During the DB Period
Description: as for outcome 6
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 62
score on scale
  Baseline | 40.72 (11.86) | 46.02 (10.58)
  Change from Baseline at Week 24: number analyzed (Participants) | 20 | 54
  Change from Baseline at Week 24 | 1.49 (10.22) | 2.33 (8.29)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 46
  Change from Baseline at Week 48 | 4.79 (9.07) | 4.15 (7.49)
  Change from Baseline at Week 72: number analyzed (Participants) | 13 | 43
  Change from Baseline at Week 72 | 3.43 (9.38) | 3.68 (6.43)
  Change from Baseline at Week 96: number analyzed (Participants) | 8 | 31
  Change from Baseline at Week 96 | 0.00 (7.94) | 4.34 (9.39)
  Change from Baseline at Week 120: number analyzed (Participants) | 3 | 16
  Change from Baseline at Week 120 | -1.98 (11.24) | 3.96 (9.94)
  Change from Baseline at Week 144: number analyzed (Participants) | 2 | 12
  Change from Baseline at Week 144 | -9.41 (7.70) | 4.95 (7.95)
  Change from Baseline at Week 168: number analyzed (Participants) | 1 | 10
  Change from Baseline at Week 168 | -5.94 (NA) — SD was not calculable for 1 participant. | 5.05 (6.58)
  Change from Baseline at Week 192: number analyzed (Participants) | 1 | 2
  Change from Baseline at Week 192 | -11.88 (NA) — SD was not calculable for 1 participant. | 0.00 (8.40)
  Change from Baseline at Week 216: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 216 | -11.88 (NA) — SD was not calculable for 1 participant. |

14. Secondary Outcome: Change From Baseline in SF-36 Mental Component Summary Scores at 24 Week Intervals During the DB Period
Description: The SF-36v2 is a multi-purpose, short form health survey with 36 questions. It has 8 domains (vitality, physical functioning, bodily pain, general health, role-physical, role emotional, social role functioning and mental health) of functional health and well-being scores as well as psychometrically based physical and mental health summary measures and a preference-based health utility index. The component scores were transformed to a 0-100 scale, where higher score indicates better quality of life. A positive change from baseline indicates an improvement.
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 62
score on scale
  Baseline | 44.03 (13.93) | 46.43 (11.55)
  Change from Baseline at Week 24: number analyzed (Participants) | 20 | 54
  Change from Baseline at Week 24 | -0.28 (11.19) | 2.89 (8.96)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 46
  Change from Baseline at Week 48 | 0.09 (8.96) | 2.63 (8.04)
  Change from Baseline at Week 72: number analyzed (Participants) | 13 | 43
  Change from Baseline at Week 72 | 1.54 (8.18) | 3.17 (7.70)
  Change from Baseline at Week 96: number analyzed (Participants) | 8 | 31
  Change from Baseline at Week 96 | -2.65 (6.05) | 1.91 (9.32)
  Change from Baseline at Week 120: number analyzed (Participants) | 3 | 16
  Change from Baseline at Week 120 | -10.65 (11.99) | 1.03 (12.92)
  Change from Baseline at Week 144: number analyzed (Participants) | 2 | 12
  Change from Baseline at Week 144 | -5.40 (8.41) | 2.98 (12.99)
  Change from Baseline at Week 168: number analyzed (Participants) | 1 | 10
  Change from Baseline at Week 168 | -0.61 (NA) — SD was not calculable for 1 participant. | 1.63 (11.86)
  Change from Baseline at Week 192: number analyzed (Participants) | 1 | 2
  Change from Baseline at Week 192 | -14.38 (NA) — SD was not calculable for 1 participant. | -5.88 (7.54)
  Change from Baseline at Week 216: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 216 | -4.22 (NA) — SD was not calculable for 1 participant. |

15. Secondary Outcome: Change From Baseline in SF-36 Physical Component Summary Scores at 24 Week Intervals During the DB Period
Description: as for outcome 14
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 62
score on scale
  Baseline | 38.89 (11.20) | 38.59 (9.68)
  Change from Baseline at Week 24: number analyzed (Participants) | 20 | 54
  Change from Baseline at Week 24 | 1.78 (4.99) | 1.05 (6.14)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 46
  Change from Baseline at Week 48 | 3.57 (4.94) | 2.85 (4.90)
  Change from Baseline at Week 72: number analyzed (Participants) | 13 | 43
  Change from Baseline at Week 72 | 5.68 (7.32) | 2.87 (6.80)
  Change from Baseline at Week 96: number analyzed (Participants) | 8 | 31
  Change from Baseline at Week 96 | 7.25 (7.08) | 4.20 (5.90)
  Change from Baseline at Week 120: number analyzed (Participants) | 3 | 16
  Change from Baseline at Week 120 | 8.95 (8.51) | 2.68 (8.72)
  Change from Baseline at Week 144: number analyzed (Participants) | 2 | 12
  Change from Baseline at Week 144 | 3.18 (10.67) | 2.89 (7.11)
  Change from Baseline at Week 168: number analyzed (Participants) | 1 | 10
  Change from Baseline at Week 168 | -2.00 (NA) — SD was not calculable for 1 participant. | 1.83 (10.96)
  Change from Baseline at Week 192: number analyzed (Participants) | 1 | 2
  Change from Baseline at Week 192 | -1.79 (NA) — SD was not calculable for 1 participant. | 7.24 (3.35)
  Change from Baseline at Week 216: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 216 | -10.84 (NA) — SD was not calculable for 1 participant. |

16. Secondary Outcome: Change From Baseline in EuroQoL-5 Dimensions (EQ-5D) Index Scores at 24 Week Intervals During the DB Period
Description: The EQ-5D is a participant-answered questionnaire measuring 5 dimensions of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression with 3 possible response categories: 1) no problems; 2) some problems; 3) severe problems. The scores from 5 dimensions are used as input to generate EQ-5D index score using scoring algorithm. The EQ-5D index score is scored on a scale of -0.2 to 1. A higher score reflects a better health state. A positive change from baseline indicates an improvement
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 62
score on scale
  Baseline | 0.7153 (0.2253) | 0.6881 (0.2040)
  Change from Baseline at Week 24: number analyzed (Participants) | 20 | 53
  Change from Baseline at Week 24 | 0.0031 (0.1602) | 0.0188 (0.1812)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 45
  Change from Baseline at Week 48 | 0.0016 (0.1176) | 0.0244 (0.1571)
  Change from Baseline at Week 72: number analyzed (Participants) | 12 | 42
  Change from Baseline at Week 72 | 0.0582 (0.1498) | 0.0238 (0.1323)
  Change from Baseline at Week 96: number analyzed (Participants) | 8 | 30
  Change from Baseline at Week 96 | 0.0447 (0.1508) | 0.0460 (0.1067)
  Change from Baseline at Week 120: number analyzed (Participants) | 3 | 16
  Change from Baseline at Week 120 | -0.0288 (0.1908) | 0.0099 (0.1636)
  Change from Baseline at Week 144: number analyzed (Participants) | 2 | 12
  Change from Baseline at Week 144 | -0.1001 (0.1416) | 0.0063 (0.2299)
  Change from Baseline at Week 168: number analyzed (Participants) | 1 | 10
  Change from Baseline at Week 168 | 0.0000 (NA) — SD was not calculable for 1 participant. | -0.0261 (0.2532)
  Change from Baseline at Week 192: number analyzed (Participants) | 1 | 2
  Change from Baseline at Week 192 | -0.2002 (NA) — SD was not calculable for 1 participant. | 0.0299 (0.0423)
  Change from Baseline at Week 216: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 216 | -0.2002 (NA) — SD was not calculable for 1 participant. |

17. Secondary Outcome: Change From Baseline in Speed of Timed 25-Foot Walk (T25W) at 24 Week Intervals During the DB Period
Description: The T25W is an assessment of walking ability. The time (in seconds) that the participant took to walk 25 feet was measured. Speed is calculated as 1/Timed 25-Foot Walk where time is measured in seconds. A positive change from baseline indicates an improvement.
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 1/seconds
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 29 | 63
1/seconds
  Baseline | 0.1442 (0.0793) | 0.1355 (0.0561)
  Change from Baseline at Week 24: number analyzed (Participants) | 19 | 53
  Change from Baseline at Week 24 | 0.0030 (0.0374) | 0.0040 (0.0225)
  Change from Baseline at Week 48: number analyzed (Participants) | 16 | 45
  Change from Baseline at Week 48 | 0.0142 (0.0493) | 0.0115 (0.0306)
  Change from Baseline at Week 72: number analyzed (Participants) | 11 | 43
  Change from Baseline at Week 72 | 0.0205 (0.0531) | 0.0071 (0.0257)
  Change from Baseline at Week 96: number analyzed (Participants) | 6 | 31
  Change from Baseline at Week 96 | -0.0031 (0.0251) | 0.0081 (0.0253)
  Change from Baseline at Week 120: number analyzed (Participants) | 3 | 16
  Change from Baseline at Week 120 | 0.0489 (0.0301) | 0.0063 (0.0386)
  Change from Baseline at Week 144: number analyzed (Participants) | 2 | 12
  Change from Baseline at Week 144 | 0.0388 (0.0572) | 0.0003 (0.0443)
  Change from Baseline at Week 168: number analyzed (Participants) | 1 | 9
  Change from Baseline at Week 168 | -0.0656 (NA) — SD was not calculable for 1 participant. | -0.0155 (0.0379)
  Change from Baseline at Week 192: number analyzed (Participants) | 1 | 2
  Change from Baseline at Week 192 | -0.0812 (NA) — SD was not calculable for 1 participant. | -0.0304 (0.0360)
  Change from Baseline at Week 216: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 216 | -0.0917 (NA) — SD was not calculable for 1 participant. |

18. Secondary Outcome: Change From Baseline in Modified Rankin Scale (mRS) Scores at 24 Week Intervals During the DB Period
Description: The mRS is a 7-point disability scale that assesses the degree of disability in participants with neurological impairment. Possible scores range from 0 (no symptoms at all) up to 6 (death). Higher scores reflect increased disability. A negative change from baseline indicates an improvement.
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 63
score on scale
  Baseline | 1.66 (1.00) | 1.97 (0.98)
  Change from Baseline at Week 24: number analyzed (Participants) | 19 | 54
  Change from Baseline at Week 24 | -0.05 (0.40) | -0.04 (0.64)
  Change from Baseline at Week 48: number analyzed (Participants) | 17 | 46
  Change from Baseline at Week 48 | 0.00 (0.94) | -0.13 (0.78)
  Change from Baseline at Week 72: number analyzed (Participants) | 13 | 43
  Change from Baseline at Week 72 | -0.08 (1.04) | -0.12 (0.63)
  Change from Baseline at Week 96: number analyzed (Participants) | 8 | 31
  Change from Baseline at Week 96 | -0.38 (0.74) | -0.42 (0.99)
  Change from Baseline at Week 120: number analyzed (Participants) | 3 | 16
  Change from Baseline at Week 120 | -1.00 (0.00) | -0.13 (0.81)
  Change from Baseline at Week 144: number analyzed (Participants) | 2 | 11
  Change from Baseline at Week 144 | -1.00 (1.41) | -0.09 (0.54)
  Change from Baseline at Week 168: number analyzed (Participants) | 0 | 10
  Change from Baseline at Week 168 |  | 0.00 (0.67)
  Change from Baseline at Week 192: number analyzed (Participants) | 1 | 2
  Change from Baseline at Week 192 | -1.00 (NA) — SD was not calculable for 1 participant. | -0.50 (2.12)
  Change from Baseline at Week 216: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 216 | -1.00 (NA) — SD was not calculable for 1 participant. |

19. Secondary Outcome: Change From Baseline in Zarit Burden Interview (ZBI) Scores at 24 Week Intervals During the DB Period
Description: The ZBI is the measurement to assess caregiver burden. The 22 items ask for the strain caregivers perceive. Responses range from 0 (never) to 4 (nearly always). The overall ZBI score ranges from 0 to 88. The higher the total score, the heavier the perceived burden. A negative change from baseline indicates an improvement.
Time Frame: Baseline up to Week 120
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 7 | 8
score on scale
  Baseline | 19.43 (12.19) | 11.32 (7.20)
  Change from Baseline at Week 24: number analyzed (Participants) | 6 | 4
  Change from Baseline at Week 24 | 0.00 (6.20) | 1.50 (9.68)
  Change from Baseline at Week 48: number analyzed (Participants) | 6 | 2
  Change from Baseline at Week 48 | -2.83 (6.11) | -3.00 (9.90)
  Change from Baseline at Week 72: number analyzed (Participants) | 3 | 1
  Change from Baseline at Week 72 | -5.00 (3.00) | -13.00 (NA) — SD was not calculable for 1 participant.
  Change from Baseline at Week 96: number analyzed (Participants) | 2 | 0
  Change from Baseline at Week 96 | -1.00 (7.07) |
  Change from Baseline at Week 120: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 120 | 4.00 (NA) — SD was not calculable for 1 participant. |

20. Secondary Outcome: Change From Baseline in Expanded Disability Status Scale (EDSS) Scores at 24 Week Intervals During the DB Period
Description: The EDSS is an ordinal scale with values from 0 points (normal neurological examination) to 10 points (death) increasing in half-point increments once an EDSS of 1.0 has been reached. Higher scores represent increased disability. A negative change from baseline indicates an improvement.
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 63
score on scale
  Baseline | 3.66 (1.61) | 3.92 (1.50)
  Change from Baseline at Week 24: number analyzed (Participants) | 20 | 53
  Change from Baseline at Week 24 | -0.03 (0.38) | -0.24 (0.71)
  Change from Baseline at Week 48: number analyzed (Participants) | 18 | 46
  Change from Baseline at Week 48 | -0.06 (0.42) | -0.32 (0.65)
  Change from Baseline at Week 72: number analyzed (Participants) | 12 | 42
  Change from Baseline at Week 72 | 0.21 (0.58) | -0.29 (0.76)
  Change from Baseline at Week 96: number analyzed (Participants) | 8 | 29
  Change from Baseline at Week 96 | -0.50 (0.76) | -0.03 (0.48)
  Change from Baseline at Week 120: number analyzed (Participants) | 3 | 16
  Change from Baseline at Week 120 | -0.50 (0.87) | -0.22 (0.91)
  Change from Baseline at Week 144: number analyzed (Participants) | 2 | 11
  Change from Baseline at Week 144 | -1.00 (0.71) | 0.18 (0.68)
  Change from Baseline at Week 168: number analyzed (Participants) | 1 | 10
  Change from Baseline at Week 168 | -0.50 (NA) — SD was not calculable for 1 participant. | -0.15 (1.13)
  Change from Baseline at Week 192: number analyzed (Participants) | 1 | 2
  Change from Baseline at Week 192 | 0.00 (NA) — SD was not calculable for 1 participant. | 0.25 (1.06)
  Change from Baseline at Week 216: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 216 | -0.50 (NA) — SD was not calculable for 1 participant. |

21. Secondary Outcome: Change From Baseline in Visual Acuity (Snellen Chart) at 24 Week Intervals During the DB Period
Description: Visual acuity was measured using Snellen 20-foot wall chart and then converted to logMAR visual acuity scoring. Lower values indicate better visual acuity. Data are reported for right eye (OD) and left eye (OS). A negative change from baseline indicates an improvement.
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: LogMAR units
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 63
LogMAR units
  Baseline: OD | 0.560 (0.903) | 0.449 (0.712)
  Baseline: OS | 0.456 (0.811) | 0.545 (0.836)
  Change from Baseline at Week 24: OD: number analyzed (Participants) | 20 | 53
  Change from Baseline at Week 24: OD | -0.058 (0.512) | 0.039 (0.434)
  Change from Baseline at Week 24: OS: number analyzed (Participants) | 20 | 53
  Change from Baseline at Week 24: OS | 0.046 (0.242) | -0.001 (0.500)
  Change from Baseline at Week 48: OD: number analyzed (Participants) | 18 | 46
  Change from Baseline at Week 48: OD | -0.027 (0.097) | 0.053 (0.434)
  Change from Baseline at Week 48: OS: number analyzed (Participants) | 18 | 46
  Change from Baseline at Week 48: OS | 0.050 (0.252) | -0.006 (0.591)
  Change from Baseline at Week 72: OD: number analyzed (Participants) | 12 | 42
  Change from Baseline at Week 72: OD | -0.050 (0.140) | -0.056 (0.260)
  Change from Baseline at Week 72: OS: number analyzed (Participants) | 12 | 42
  Change from Baseline at Week 72: OS | -0.083 (0.595) | -0.101 (0.492)
  Change from Baseline at Week 96: OD: number analyzed (Participants) | 8 | 29
  Change from Baseline at Week 96: OD | -0.045 (0.099) | -0.081 (0.580)
  Change from Baseline at Week 96: OS: number analyzed (Participants) | 8 | 29
  Change from Baseline at Week 96: OS | -0.260 (0.707) | -0.121 (0.571)
  Change from Baseline at Week 120: OD: number analyzed (Participants) | 3 | 16
  Change from Baseline at Week 120: OD | -0.027 (0.142) | -0.039 (0.637)
  Change from Baseline at Week 120: OS: number analyzed (Participants) | 3 | 15
  Change from Baseline at Week 120: OS | 0.000 (0.000) | -0.229 (0.754)
  Change from Baseline at Week 144: OD: number analyzed (Participants) | 2 | 11
  Change from Baseline at Week 144: OD | 0.010 (0.127) | 0.149 (0.618)
  Change from Baseline at Week 144: OS: number analyzed (Participants) | 2 | 11
  Change from Baseline at Week 144: OS | 0.000 (0.000) | -0.280 (0.846)
  Change from Baseline at Week 168: OD: number analyzed (Participants) | 1 | 10
  Change from Baseline at Week 168: OD | -0.080 (NA) — SD was not calculable for 1 participant. | 0.134 (0.663)
  Change from Baseline at Week 168: OS: number analyzed (Participants) | 1 | 10
  Change from Baseline at Week 168: OS | -0.100 (NA) — SD was not calculable for 1 participant. | -0.320 (0.910)
  Change from Baseline at Week 192: OD: number analyzed (Participants) | 1 | 2
  Change from Baseline at Week 192: OD | -0.180 (NA) — SD was not calculable for 1 participant. | -0.110 (0.156)
  Change from Baseline at Week 192: OS: number analyzed (Participants) | 1 | 2
  Change from Baseline at Week 192: OS | 0.080 (NA) — SD was not calculable for 1 participant. | -0.050 (0.071)
  Change from Baseline at Week 216: OD: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 216: OD | -0.180 (NA) — SD was not calculable for 1 participant. |
  Change from Baseline at Week 216: OS: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 216: OS | -0.100 (NA) — SD was not calculable for 1 participant. |

22. Secondary Outcome: Change From Baseline in Visual Function (Low-Contrast Sloan Letter Chart [LCSLC]) Scores at 24 Week Intervals During the DB Period
Description: The LCSLC evaluates the visual function and captures the minimum size at which individuals can perceive letters of a particular contrast level. The change in binocular visual acuity, as assessed by the number of letters read correctly from a distance of 2 meters on 100%, 2.5% and 1.25% contrast level Sloan letter charts, was analyzed. The LCSLC is scored on a scale of 0-60. Higher scores indicate better visual function. A positive change from baseline indicates an improvement.
Time Frame: Baseline up to Week 216
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 29 | 60
letters
  Baseline: 100% CHART | 44.3 (16.1) | 44.4 (16.3)
  Baseline: 2.5% CHART | 24.6 (16.2) | 22.6 (15.6)
  Baseline: 1.25% CHART | 17.5 (15.7) | 14.9 (14.8)
  Change from Baseline at Week 24: 100% CHART: number analyzed (Participants) | 19 | 49
  Change from Baseline at Week 24: 100% CHART | 0.5 (7.1) | 2.0 (5.3)
  Change from Baseline at Week 24: 2.5% CHART: number analyzed (Participants) | 19 | 49
  Change from Baseline at Week 24: 2.5% CHART | -2.8 (9.1) | 1.7 (7.1)
  Change from Baseline at Week 24: 1.25% CHART: number analyzed (Participants) | 19 | 49
  Change from Baseline at Week 24: 1.25% CHART | -4.2 (11.9) | 0.1 (7.5)
  Change from Baseline at Week 48: 100% CHART: number analyzed (Participants) | 16 | 43
  Change from Baseline at Week 48: 100% CHART | -3.4 (8.7) | 1.3 (6.1)
  Change from Baseline at Week 48: 2.5% CHART: number analyzed (Participants) | 15 | 43
  Change from Baseline at Week 48: 2.5% CHART | 1.5 (6.1) | 4.0 (9.2)
  Change from Baseline at Week 48: 1.25% CHART: number analyzed (Participants) | 15 | 43
  Change from Baseline at Week 48: 1.25% CHART | 1.7 (11.3) | 4.1 (9.3)
  Change from Baseline at Week 72: 100% CHART: number analyzed (Participants) | 11 | 41
  Change from Baseline at Week 72: 100% CHART | 0.3 (5.9) | 2.8 (7.3)
  Change from Baseline at Week 72: 2.5% CHART: number analyzed (Participants) | 11 | 41
  Change from Baseline at Week 72: 2.5% CHART | -0.6 (8.6) | 2.6 (7.5)
  Change from Baseline at Week 72: 1.25% CHART: number analyzed (Participants) | 11 | 41
  Change from Baseline at Week 72: 1.25% CHART | -2.4 (8.3) | 0.4 (10.6)
  Change from Baseline at Week 96: 100% CHART: number analyzed (Participants) | 7 | 28
  Change from Baseline at Week 96: 100% CHART | 3.3 (13.2) | 2.1 (12.4)
  Change from Baseline at Week 96: 2.5% CHART: number analyzed (Participants) | 7 | 28
  Change from Baseline at Week 96: 2.5% CHART | 2.6 (20.1) | 2.3 (10.8)
  Change from Baseline at Week 96: 1.25% CHART: number analyzed (Participants) | 7 | 28
  Change from Baseline at Week 96: 1.25% CHART | -3.4 (11.3) | -0.5 (11.3)
  Change from Baseline at Week 120: 100% CHART: number analyzed (Participants) | 3 | 14
  Change from Baseline at Week 120: 100% CHART | -1.0 (1.0) | 1.5 (10.6)
  Change from Baseline at Week 120: 2.5% CHART: number analyzed (Participants) | 3 | 14
  Change from Baseline at Week 120: 2.5% CHART | 3.7 (4.6) | 2.1 (7.3)
  Change from Baseline at Week 120: 1.25% CHART: number analyzed (Participants) | 3 | 14
  Change from Baseline at Week 120: 1.25% CHART | -2.0 (5.0) | 1.6 (9.1)
  Change from Baseline at Week 144: 100% CHART: number analyzed (Participants) | 2 | 10
  Change from Baseline at Week 144: 100% CHART | -3.5 (2.1) | 0.4 (7.7)
  Change from Baseline at Week 144: 2.5% CHART: number analyzed (Participants) | 2 | 10
  Change from Baseline at Week 144: 2.5% CHART | 17.5 (17.7) | 1.6 (12.0)
  Change from Baseline at Week 144: 1.25% CHART: number analyzed (Participants) | 2 | 10
  Change from Baseline at Week 144: 1.25% CHART | -7.0 (7.1) | 1.4 (12.2)
  Change from Baseline at Week 168: 100% CHART: number analyzed (Participants) | 0 | 10
  Change from Baseline at Week 168: 100% CHART |  | 2.1 (6.7)
  Change from Baseline at Week 168: 2.5% CHART: number analyzed (Participants) | 0 | 10
  Change from Baseline at Week 168: 2.5% CHART |  | 6.2 (8.2)
  Change from Baseline at Week 168: 1.25% CHART: number analyzed (Participants) | 0 | 10
  Change from Baseline at Week 168: 1.25% CHART |  | 0.3 (12.2)
  Change from Baseline at Week 192: 100% CHART: number analyzed (Participants) | 1 | 2
  Change from Baseline at Week 192: 100% CHART | 1.0 (NA) — SD was not calculable for 1 participant. | -2.5 (3.5)
  Change from Baseline at Week 192: 2.5% CHART: number analyzed (Participants) | 1 | 2
  Change from Baseline at Week 192: 2.5% CHART | -1.0 (NA) — SD was not calculable for 1 participant. | -1.0 (4.2)
  Change from Baseline at Week 192: 1.25% CHART: number analyzed (Participants) | 1 | 2
  Change from Baseline at Week 192: 1.25% CHART | -8.0 (NA) — SD was not calculable for 1 participant. | -4.0 (7.1)
  Change from Baseline at Week 216: 100% CHART: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 216: 100% CHART | 0.0 (NA) — SD was not calculable for 1 participant. |
  Change from Baseline at Week 216: 2.5% CHART: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 216: 2.5% CHART | -1.0 (NA) — SD was not calculable for 1 participant. |
  Change from Baseline at Week 216: 1.25% CHART: number analyzed (Participants) | 1 | 0
  Change from Baseline at Week 216: 1.25% CHART | -8.0 (NA) — SD was not calculable for 1 participant. |

23. Secondary Outcome: Number of Participants With at Least One Adverse Event in the DB Period
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Pre-existing conditions which worsen during a study are also considered as adverse events.
Time Frame: Up to Week 216
Population: The Safety Analysis Population (SAF) included all randomized participants who had received at least 1 dose of satralizumab or placebo.
Measure: Number; unit: participants
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 63
participants | 24 | 58

24. Secondary Outcome: Number of Participants With at Least One Serious Adverse Event in the DB Period
Description: A serious adverse event is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, or is medically significant or requires intervention to prevent one or other of the outcomes listed above.
Time Frame: Up to Week 216
Population: The SAF included all randomized participants who had received at least 1 dose of satralizumab or placebo.
Measure: Number; unit: participants
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 63
participants | 5 | 12

25. Secondary Outcome: Number of Participants With Non-Serious Adverse Events of Special Interest in the DB Period
Description: Non-serious adverse events of special interest for this study included:
  1) cases of an elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) in combination with either an elevated bilirubin or clinical jaundice, 2) suspected transmission of an infectious agent by the study treatment.
Time Frame: Up to Week 216
Population: The SAF included all randomized participants who had received at least 1 dose of satralizumab or placebo.
Measure: Number; unit: participants
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 63
participants | 0 | 0

26. Secondary Outcome: Number of Participants With Selected Adverse Events in the DB Period
Description: Selected adverse events for this study included:
  1) all infections, 2) serious infections, 3) potential opportunistic infections, 4) injection-related reactions (IRRs; an AE which occured within 24 hours after study treatment injection except where the event was not considered an allergic reaction), 5) psychiatric disorders and 6) anaphylaxis (an acute allergic/hypersensitivity reaction).
Time Frame: Up to Week 216
Population: The SAF included all randomized participants who had received at least 1 dose of satralizumab or placebo.
Measure: Number; unit: participants
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 63
participants
  All Infections | 14 | 34
  Serious Infections | 3 | 6
  Potential Opportunistic Infections | 5 | 3
  Injection-related Reactions | 5 | 8
  Psychiatric Disorders | 4 | 13
  Anaphylaxis | 0 | 0

27. Secondary Outcome: Number of Participants With Suicidal Behaviors and Ideations Collected by Columbia-Suicide Severity Rating Scale in the DB Period
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS) is an assessment tool to evaluate suicidal ideation and behavior. Categories have binary responses (yes/no) and include: Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent, Preparatory Acts and Behavior; Aborted Attempt; Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide. Suicidal ideation or behavior is indicated by a "yes" answer to any of the listed categories. A score of 0 is assigned if no suicide risk is present. A score of 1 or higher indicates suicidal ideation or behavior.
Time Frame: Baseline and Post-Baseline (up to Week 216)
Population: The SAF included all randomized participants who had received at least 1 dose of satralizumab or placebo.
Measure: Number; unit: participants
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 63
participants
  Baseline | 0 | 9
  Post-Baseline | 1 | 3

28. Secondary Outcome: Serum Satralizumab Concentration During the DB Period
Time Frame: Baseline, Weeks 2, 4, 5, 6, 8, and every 4 weeks thereafter up to Week 204
Population: Participants from SAF who received satralizumab were evaluated for this outcome measure. The SAF included all randomized participants who had received at least 1 dose of satralizumab or placebo. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 62
ng/mL
  Baseline | 145.13 (274.87)
  Week 2: number analyzed (Participants) | 61
  Week 2 | 8099.70 (4541.66)
  Week 4: number analyzed (Participants) | 56
  Week 4 | 14602.50 (8931.85)
  Week 5: number analyzed (Participants) | 44
  Week 5 | 22564.32 (12306.09)
  Week 6: number analyzed (Participants) | 42
  Week 6 | 20991.43 (12515.82)
  Week 8: number analyzed (Participants) | 60
  Week 8 | 14864.35 (9955.41)
  Week 12: number analyzed (Participants) | 55
  Week 12 | 14760.33 (10695.11)
  Week 16: number analyzed (Participants) | 53
  Week 16 | 14613.11 (11276.95)
  Week 20: number analyzed (Participants) | 55
  Week 20 | 14136.62 (12489.83)
  Week 24: number analyzed (Participants) | 55
  Week 24 | 15634.18 (13310.22)
  Week 28: number analyzed (Participants) | 53
  Week 28 | 15538.38 (13406.73)
  Week 32: number analyzed (Participants) | 52
  Week 32 | 15111.94 (13827.06)
  Week 36: number analyzed (Participants) | 50
  Week 36 | 16068.58 (14643.61)
  Week 40: number analyzed (Participants) | 46
  Week 40 | 15428.04 (16059.35)
  Week 44: number analyzed (Participants) | 46
  Week 44 | 16110.00 (15363.29)
  Week 48: number analyzed (Participants) | 44
  Week 48 | 16701.16 (16790.77)
  Week 52: number analyzed (Participants) | 44
  Week 52 | 15300.57 (14701.05)
  Week 56: number analyzed (Participants) | 45
  Week 56 | 16390.82 (16130.69)
  Week 60: number analyzed (Participants) | 43
  Week 60 | 16050.81 (14779.35)
  Week 64: number analyzed (Participants) | 42
  Week 64 | 14385.10 (14084.24)
  Week 68: number analyzed (Participants) | 41
  Week 68 | 14010.46 (13614.03)
  Week 72: number analyzed (Participants) | 42
  Week 72 | 12895.69 (13849.12)
  Week 76: number analyzed (Participants) | 42
  Week 76 | 14139.31 (14549.71)
  Week 80: number analyzed (Participants) | 42
  Week 80 | 12709.79 (14098.26)
  Week 84: number analyzed (Participants) | 40
  Week 84 | 11725.05 (13654.04)
  Week 88: number analyzed (Participants) | 35
  Week 88 | 13733.17 (13438.07)
  Week 92: number analyzed (Participants) | 32
  Week 92 | 12928.13 (13302.53)
  Week 96: number analyzed (Participants) | 31
  Week 96 | 14036.58 (12644.16)
  Week 100: number analyzed (Participants) | 20
  Week 100 | 14186.50 (12888.23)
  Week 104: number analyzed (Participants) | 22
  Week 104 | 16647.00 (15568.61)
  Week 108: number analyzed (Participants) | 22
  Week 108 | 15970.00 (13525.53)
  Week 112: number analyzed (Participants) | 19
  Week 112 | 18657.37 (17426.82)
  Week 116: number analyzed (Participants) | 15
  Week 116 | 17677.33 (16892.59)
  Week 120: number analyzed (Participants) | 14
  Week 120 | 16615.00 (16751.13)
  Week 124: number analyzed (Participants) | 15
  Week 124 | 13734.00 (12687.75)
  Week 128: number analyzed (Participants) | 15
  Week 128 | 13738.00 (16005.33)
  Week 132: number analyzed (Participants) | 15
  Week 132 | 13311.73 (15401.04)
  Week 136: number analyzed (Participants) | 13
  Week 136 | 14208.54 (15266.48)
  Week 140: number analyzed (Participants) | 13
  Week 140 | 13404.62 (12392.48)
  Week 144: number analyzed (Participants) | 11
  Week 144 | 16138.18 (13782.26)
  Week 148: number analyzed (Participants) | 12
  Week 148 | 14044.33 (12082.37)
  Week 152: number analyzed (Participants) | 12
  Week 152 | 14644.42 (13123.67)
  Week 156: number analyzed (Participants) | 11
  Week 156 | 18856.36 (20378.31)
  Week 160: number analyzed (Participants) | 11
  Week 160 | 15238.18 (11360.62)
  Week 164: number analyzed (Participants) | 11
  Week 164 | 14760.00 (11479.99)
  Week 168: number analyzed (Participants) | 10
  Week 168 | 14199.60 (9911.22)
  Week 172: number analyzed (Participants) | 7
  Week 172 | 17971.43 (16962.78)
  Week 176: number analyzed (Participants) | 7
  Week 176 | 17922.86 (12815.57)
  Week 180: number analyzed (Participants) | 7
  Week 180 | 15981.43 (9640.78)
  Week 184: number analyzed (Participants) | 6
  Week 184 | 17911.67 (15142.19)
  Week 188: number analyzed (Participants) | 4
  Week 188 | 16442.50 (13180.44)
  Week 192: number analyzed (Participants) | 2
  Week 192 | 28750.00 (22415.28)
  Week 196: number analyzed (Participants) | 2
  Week 196 | 26850.00 (20152.54)
  Week 200: number analyzed (Participants) | 1
  Week 200 | 45000.00 (NA) — SD was not calculable for 1 participant.
  Week 204: number analyzed (Participants) | 1
  Week 204 | 34500.00 (NA) — SD was not calculable for 1 participant.

29. Secondary Outcome: Serum Interleukin-6 (IL-6) Concentration During the DB Period
Time Frame: Baseline, Weeks 2, 4, and every 4 weeks thereafter up to Week 216
Population: The SAF included all randomized participants who had received at least 1 dose of satralizumab or placebo. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 30 | 62
pg/mL
  Baseline: number analyzed (Participants) | 29 | 62
  Baseline | 3.66 (6.49) | 3.49 (5.14)
  Week 2: number analyzed (Participants) | 30 | 60
  Week 2 | 5.90 (16.31) | 30.14 (26.07)
  Week 4: number analyzed (Participants) | 28 | 61
  Week 4 | 5.41 (10.02) | 51.53 (126.49)
  Week 8: number analyzed (Participants) | 26 | 61
  Week 8 | 3.30 (4.59) | 30.88 (25.57)
  Week 12: number analyzed (Participants) | 25 | 53
  Week 12 | 3.40 (4.21) | 32.02 (24.91)
  Week 16: number analyzed (Participants) | 23 | 53
  Week 16 | 3.72 (4.54) | 28.59 (23.27)
  Week 20: number analyzed (Participants) | 22 | 55
  Week 20 | 2.99 (2.88) | 24.06 (19.59)
  Week 24: number analyzed (Participants) | 20 | 55
  Week 24 | 3.68 (4.02) | 26.27 (23.19)
  Week 28: number analyzed (Participants) | 20 | 53
  Week 28 | 3.88 (4.24) | 26.89 (24.01)
  Week 32: number analyzed (Participants) | 22 | 52
  Week 32 | 3.43 (3.20) | 33.29 (37.93)
  Week 36: number analyzed (Participants) | 20 | 50
  Week 36 | 3.78 (3.65) | 26.03 (21.75)
  Week 40: number analyzed (Participants) | 19 | 46
  Week 40 | 4.82 (6.45) | 24.16 (19.93)
  Week 44: number analyzed (Participants) | 18 | 46
  Week 44 | 3.47 (3.65) | 26.16 (20.39)
  Week 48: number analyzed (Participants) | 17 | 43
  Week 48 | 4.58 (4.21) | 29.61 (27.37)
  Week 52: number analyzed (Participants) | 18 | 44
  Week 52 | 3.52 (3.36) | 26.94 (22.26)
  Week 56: number analyzed (Participants) | 15 | 45
  Week 56 | 4.13 (5.26) | 33.15 (40.66)
  Week 60: number analyzed (Participants) | 12 | 43
  Week 60 | 3.28 (3.65) | 31.34 (25.38)
  Week 64: number analyzed (Participants) | 14 | 41
  Week 64 | 4.08 (4.48) | 30.60 (24.55)
  Week 68: number analyzed (Participants) | 14 | 41
  Week 68 | 2.75 (3.35) | 30.56 (44.67)
  Week 72: number analyzed (Participants) | 12 | 41
  Week 72 | 2.95 (4.80) | 23.16 (17.54)
  Week 76: number analyzed (Participants) | 12 | 42
  Week 76 | 2.44 (3.04) | 24.08 (16.78)
  Week 80: number analyzed (Participants) | 11 | 41
  Week 80 | 1.57 (0.00) | 24.86 (17.89)
  Week 84: number analyzed (Participants) | 12 | 40
  Week 84 | 2.27 (1.84) | 27.61 (23.04)
  Week 88: number analyzed (Participants) | 9 | 35
  Week 88 | 1.57 (0.00) | 26.51 (20.07)
  Week 92: number analyzed (Participants) | 10 | 31
  Week 92 | 3.38 (4.80) | 25.48 (17.24)
  Week 96: number analyzed (Participants) | 7 | 31
  Week 96 | 1.57 (0.00) | 24.57 (15.25)
  Week 100: number analyzed (Participants) | 5 | 18
  Week 100 | 1.57 (0.00) | 26.31 (18.74)
  Week 104: number analyzed (Participants) | 7 | 22
  Week 104 | 1.57 (0.00) | 26.30 (19.96)
  Week 108: number analyzed (Participants) | 6 | 21
  Week 108 | 1.57 (0.00) | 27.64 (23.97)
  Week 112: number analyzed (Participants) | 3 | 19
  Week 112 | 1.57 (0.00) | 27.39 (22.72)
  Week 116: number analyzed (Participants) | 4 | 15
  Week 116 | 1.57 (0.00) | 31.73 (23.27)
  Week 120: number analyzed (Participants) | 3 | 13
  Week 120 | 1.57 (0.00) | 55.92 (68.46)
  Week 124: number analyzed (Participants) | 3 | 15
  Week 124 | 1.57 (0.00) | 29.46 (19.49)
  Week 128: number analyzed (Participants) | 2 | 14
  Week 128 | 1.57 (0.00) | 31.20 (21.29)
  Week 132: number analyzed (Participants) | 2 | 15
  Week 132 | 1.57 (0.00) | 33.84 (34.36)
  Week 136: number analyzed (Participants) | 2 | 13
  Week 136 | 1.57 (0.00) | 51.83 (73.68)
  Week 140: number analyzed (Participants) | 1 | 12
  Week 140 | 1.57 (NA) — SD was not calculable for 1 participant. | 41.00 (45.44)
  Week 144: number analyzed (Participants) | 2 | 11
  Week 144 | 1.57 (0.00) | 28.26 (25.64)
  Week 148: number analyzed (Participants) | 2 | 12
  Week 148 | 1.57 (0.00) | 28.76 (21.52)
  Week 152: number analyzed (Participants) | 1 | 12
  Week 152 | 1.57 (NA) — SD was not calculable for 1 participant. | 28.07 (23.66)
  Week 156: number analyzed (Participants) | 1 | 11
  Week 156 | 1.57 (NA) — SD was not calculable for 1 participant. | 27.25 (19.19)
  Week 160: number analyzed (Participants) | 1 | 11
  Week 160 | 1.57 (NA) — SD was not calculable for 1 participant. | 29.60 (20.30)
  Week 164: number analyzed (Participants) | 1 | 11
  Week 164 | 1.57 (NA) — SD was not calculable for 1 participant. | 34.00 (24.13)
  Week 168: number analyzed (Participants) | 1 | 10
  Week 168 | 1.57 (NA) — SD was not calculable for 1 participant. | 26.29 (20.85)
  Week 172: number analyzed (Participants) | 1 | 7
  Week 172 | 1.57 (NA) — SD was not calculable for 1 participant. | 23.57 (6.59)
  Week 176: number analyzed (Participants) | 1 | 7
  Week 176 | 1.57 (NA) — SD was not calculable for 1 participant. | 27.73 (11.10)
  Week 180: number analyzed (Participants) | 1 | 7
  Week 180 | 1.57 (NA) — SD was not calculable for 1 participant. | 24.09 (9.21)
  Week 184: number analyzed (Participants) | 1 | 6
  Week 184 | 3.63 (NA) — SD was not calculable for 1 participant. | 17.34 (8.47)
  Week 188: number analyzed (Participants) | 1 | 4
  Week 188 | 5.21 (NA) — SD was not calculable for 1 participant. | 17.78 (7.22)
  Week 192: number analyzed (Participants) | 1 | 2
  Week 192 | 1.57 (NA) — SD was not calculable for 1 participant. | 16.55 (3.89)
  Week 196: number analyzed (Participants) | 1 | 2
  Week 196 | 1.57 (NA) — SD was not calculable for 1 participant. | 14.45 (2.76)
  Week 200: number analyzed (Participants) | 1 | 1
  Week 200 | 1.57 (NA) — SD was not calculable for 1 participant. | 36.90 (NA) — SD was not calculable for 1 participant.
  Week 204: number analyzed (Participants) | 1 | 1
  Week 204 | 1.57 (NA) — SD was not calculable for 1 participant. | 12.30 (NA) — SD was not calculable for 1 participant.
  Week 208: number analyzed (Participants) | 1 | 0
  Week 208 | 1.57 (NA) — SD was not calculable for 1 participant. |
  Week 212: number analyzed (Participants) | 1 | 0
  Week 212 | 1.57 (NA) — SD was not calculable for 1 participant. |
  Week 216: number analyzed (Participants) | 1 | 0
  Week 216 | 1.57 (NA) — SD was not calculable for 1 participant. |

30. Secondary Outcome: Serum Soluble IL-6 Receptor (sIL-6R) Concentration During the DB Period
Time Frame: Baseline, Weeks 2, 4, and every 4 weeks thereafter up to Week 216
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 62
ng/mL
  Baseline | 31.88 (7.50) | 33.18 (7.72)
  Week 2: number analyzed (Participants) | 30 | 61
  Week 2 | 32.72 (8.09) | 396.49 (80.09)
  Week 4: number analyzed (Participants) | 29 | 61
  Week 4 | 44.79 (64.73) | 509.21 (121.99)
  Week 8: number analyzed (Participants) | 27 | 61
  Week 8 | 33.23 (7.21) | 560.63 (164.11)
  Week 12: number analyzed (Participants) | 26 | 55
  Week 12 | 33.02 (7.65) | 582.36 (169.71)
  Week 16: number analyzed (Participants) | 24 | 53
  Week 16 | 31.60 (8.18) | 582.22 (204.20)
  Week 20: number analyzed (Participants) | 22 | 55
  Week 20 | 32.99 (8.14) | 555.64 (210.76)
  Week 24: number analyzed (Participants) | 20 | 55
  Week 24 | 32.47 (8.69) | 573.01 (217.93)
  Week 28: number analyzed (Participants) | 20 | 53
  Week 28 | 31.83 (9.71) | 565.29 (219.88)
  Week 32: number analyzed (Participants) | 22 | 52
  Week 32 | 33.33 (9.97) | 564.13 (215.59)
  Week 36: number analyzed (Participants) | 20 | 50
  Week 36 | 34.03 (7.79) | 572.31 (207.35)
  Week 40: number analyzed (Participants) | 19 | 46
  Week 40 | 33.64 (9.44) | 554.90 (241.34)
  Week 44: number analyzed (Participants) | 18 | 46
  Week 44 | 33.97 (9.05) | 585.62 (219.45)
  Week 48: number analyzed (Participants) | 17 | 44
  Week 48 | 33.72 (8.18) | 591.06 (213.04)
  Week 52: number analyzed (Participants) | 18 | 44
  Week 52 | 33.47 (7.58) | 575.56 (210.84)
  Week 56: number analyzed (Participants) | 15 | 45
  Week 56 | 30.34 (5.21) | 585.40 (233.38)
  Week 60: number analyzed (Participants) | 13 | 43
  Week 60 | 30.58 (6.81) | 586.40 (226.21)
  Week 64: number analyzed (Participants) | 14 | 42
  Week 64 | 32.27 (7.63) | 602.72 (239.25)
  Week 68: number analyzed (Participants) | 14 | 41
  Week 68 | 31.19 (7.23) | 617.80 (244.63)
  Week 72: number analyzed (Participants) | 13 | 42
  Week 72 | 31.12 (7.76) | 543.95 (224.00)
  Week 76: number analyzed (Participants) | 12 | 42
  Week 76 | 30.56 (7.06) | 558.67 (234.41)
  Week 80: number analyzed (Participants) | 11 | 41
  Week 80 | 33.36 (9.91) | 558.73 (235.60)
  Week 84: number analyzed (Participants) | 12 | 40
  Week 84 | 30.95 (8.96) | 552.37 (226.76)
  Week 88: number analyzed (Participants) | 10 | 35
  Week 88 | 32.05 (7.23) | 547.93 (211.74)
  Week 92: number analyzed (Participants) | 10 | 32
  Week 92 | 28.93 (5.72) | 580.64 (201.78)
  Week 96: number analyzed (Participants) | 8 | 31
  Week 96 | 32.88 (5.62) | 561.64 (205.00)
  Week 100: number analyzed (Participants) | 7 | 19
  Week 100 | 31.84 (7.62) | 559.18 (194.43)
  Week 104: number analyzed (Participants) | 7 | 22
  Week 104 | 31.70 (8.81) | 598.05 (192.99)
  Week 108: number analyzed (Participants) | 6 | 21
  Week 108 | 30.55 (6.94) | 592.06 (193.20)
  Week 112: number analyzed (Participants) | 4 | 19
  Week 112 | 29.93 (8.47) | 603.31 (227.68)
  Week 116: number analyzed (Participants) | 4 | 15
  Week 116 | 34.30 (13.37) | 609.37 (198.61)
  Week 120: number analyzed (Participants) | 3 | 13
  Week 120 | 38.20 (10.96) | 625.15 (229.67)
  Week 124: number analyzed (Participants) | 3 | 15
  Week 124 | 37.87 (13.59) | 580.07 (240.15)
  Week 128: number analyzed (Participants) | 2 | 15
  Week 128 | 44.50 (2.40) | 574.54 (214.94)
  Week 132: number analyzed (Participants) | 2 | 15
  Week 132 | 29.80 (8.63) | 575.40 (213.45)
  Week 136: number analyzed (Participants) | 2 | 13
  Week 136 | 29.45 (11.53) | 593.92 (209.84)
  Week 140: number analyzed (Participants) | 1 | 13
  Week 140 | 37.20 (NA) — SD was not calculable for 1 participant. | 627.32 (232.08)
  Week 144: number analyzed (Participants) | 2 | 11
  Week 144 | 31.10 (10.18) | 693.82 (239.70)
  Week 148: number analyzed (Participants) | 2 | 12
  Week 148 | 28.55 (13.08) | 690.83 (142.94)
  Week 152: number analyzed (Participants) | 1 | 12
  Week 152 | 33.60 (NA) — SD was not calculable for 1 participant. | 626.41 (229.59)
  Week 156: number analyzed (Participants) | 1 | 11
  Week 156 | 39.90 (NA) — SD was not calculable for 1 participant. | 682.82 (156.88)
  Week 160: number analyzed (Participants) | 1 | 11
  Week 160 | 45.00 (NA) — SD was not calculable for 1 participant. | 694.18 (127.92)
  Week 164: number analyzed (Participants) | 1 | 11
  Week 164 | 43.00 (NA) — SD was not calculable for 1 participant. | 696.18 (106.76)
  Week 168: number analyzed (Participants) | 1 | 10
  Week 168 | 40.60 (NA) — SD was not calculable for 1 participant. | 681.00 (122.60)
  Week 172: number analyzed (Participants) | 1 | 7
  Week 172 | 49.70 (NA) — SD was not calculable for 1 participant. | 672.71 (107.83)
  Week 176: number analyzed (Participants) | 1 | 7
  Week 176 | 45.50 (NA) — SD was not calculable for 1 participant. | 700.71 (90.64)
  Week 180: number analyzed (Participants) | 1 | 7
  Week 180 | 55.60 (NA) — SD was not calculable for 1 participant. | 702.00 (75.60)
  Week 184: number analyzed (Participants) | 1 | 6
  Week 184 | 41.60 (NA) — SD was not calculable for 1 participant. | 678.33 (78.20)
  Week 188: number analyzed (Participants) | 1 | 4
  Week 188 | 40.00 (NA) — SD was not calculable for 1 participant. | 688.75 (143.82)
  Week 192: number analyzed (Participants) | 1 | 2
  Week 192 | 43.40 (NA) — SD was not calculable for 1 participant. | 668.00 (192.33)
  Week 196: number analyzed (Participants) | 1 | 2
  Week 196 | 38.00 (NA) — SD was not calculable for 1 participant. | 630.00 (141.42)
  Week 200: number analyzed (Participants) | 1 | 1
  Week 200 | 35.80 (NA) — SD was not calculable for 1 participant. | 815.00 (NA) — SD was not calculable for 1 participant.
  Week 204: number analyzed (Participants) | 1 | 1
  Week 204 | 33.70 (NA) — SD was not calculable for 1 participant. | 783.00 (NA) — SD was not calculable for 1 participant.
  Week 208: number analyzed (Participants) | 1 | 0
  Week 208 | 35.60 (NA) — SD was not calculable for 1 participant. |
  Week 212: number analyzed (Participants) | 1 | 0
  Week 212 | 30.50 (NA) — SD was not calculable for 1 participant. |
  Week 216: number analyzed (Participants) | 1 | 0
  Week 216 | 37.60 (NA) — SD was not calculable for 1 participant. |

31. Secondary Outcome: Serum High Sensitivity C-Reactive Protein (hsCRP) Concentration During the DB Period
Time Frame: Baseline, Weeks 2, 4, and every 4 weeks thereafter up to Week 216
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo, Then Satralizumab | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 32 | 63
mg/L
  Baseline | 3.08 (3.77) | 4.95 (8.67)
  Week 2: number analyzed (Participants) | 30 | 62
  Week 2 | 3.51 (4.55) | 0.93 (2.35)
  Week 4: number analyzed (Participants) | 29 | 60
  Week 4 | 3.45 (6.24) | 0.82 (1.64)
  Week 8: number analyzed (Participants) | 27 | 61
  Week 8 | 4.56 (8.97) | 0.83 (1.99)
  Week 12: number analyzed (Participants) | 26 | 55
  Week 12 | 4.23 (7.23) | 1.23 (3.19)
  Week 16: number analyzed (Participants) | 24 | 53
  Week 16 | 5.30 (9.17) | 1.56 (4.53)
  Week 20: number analyzed (Participants) | 22 | 55
  Week 20 | 4.07 (5.20) | 1.78 (3.72)
  Week 24: number analyzed (Participants) | 19 | 55
  Week 24 | 3.53 (4.08) | 1.72 (4.05)
  Week 28: number analyzed (Participants) | 20 | 53
  Week 28 | 5.85 (9.99) | 2.35 (5.61)
  Week 32: number analyzed (Participants) | 22 | 52
  Week 32 | 3.97 (5.20) | 2.06 (4.28)
  Week 36: number analyzed (Participants) | 20 | 50
  Week 36 | 3.77 (4.40) | 1.56 (3.36)
  Week 40: number analyzed (Participants) | 18 | 45
  Week 40 | 6.77 (10.92) | 2.55 (5.53)
  Week 44: number analyzed (Participants) | 18 | 46
  Week 44 | 5.44 (8.72) | 3.31 (11.31)
  Week 48: number analyzed (Participants) | 17 | 44
  Week 48 | 4.70 (5.43) | 1.79 (3.24)
  Week 52: number analyzed (Participants) | 18 | 42
  Week 52 | 3.82 (4.75) | 1.90 (3.69)
  Week 56: number analyzed (Participants) | 15 | 45
  Week 56 | 5.33 (8.87) | 2.32 (5.44)
  Week 60: number analyzed (Participants) | 13 | 43
  Week 60 | 4.54 (5.60) | 3.20 (11.86)
  Week 64: number analyzed (Participants) | 14 | 43
  Week 64 | 3.76 (4.62) | 1.92 (3.55)
  Week 68: number analyzed (Participants) | 14 | 42
  Week 68 | 3.30 (5.11) | 3.65 (8.52)
  Week 72: number analyzed (Participants) | 13 | 42
  Week 72 | 5.07 (11.87) | 3.33 (7.30)
  Week 76: number analyzed (Participants) | 12 | 42
  Week 76 | 1.98 (2.12) | 2.79 (6.54)
  Week 80: number analyzed (Participants) | 11 | 41
  Week 80 | 1.10 (0.72) | 2.83 (7.09)
  Week 84: number analyzed (Participants) | 12 | 40
  Week 84 | 2.31 (4.66) | 3.81 (10.18)
  Week 88: number analyzed (Participants) | 10 | 35
  Week 88 | 1.94 (3.38) | 2.64 (6.56)
  Week 92: number analyzed (Participants) | 10 | 32
  Week 92 | 4.49 (10.18) | 1.94 (4.11)
  Week 96: number analyzed (Participants) | 8 | 31
  Week 96 | 1.76 (2.47) | 1.64 (3.37)
  Week 100: number analyzed (Participants) | 7 | 20
  Week 100 | 0.90 (0.87) | 1.87 (4.28)
  Week 104: number analyzed (Participants) | 7 | 22
  Week 104 | 1.13 (1.01) | 1.93 (4.43)
  Week 108: number analyzed (Participants) | 6 | 21
  Week 108 | 2.20 (3.16) | 2.56 (7.40)
  Week 112: number analyzed (Participants) | 4 | 19
  Week 112 | 2.25 (2.68) | 1.53 (2.86)
  Week 116: number analyzed (Participants) | 4 | 15
  Week 116 | 2.28 (3.41) | 1.19 (1.93)
  Week 120: number analyzed (Participants) | 2 | 14
  Week 120 | 1.55 (1.63) | 6.05 (14.33)
  Week 124: number analyzed (Participants) | 3 | 15
  Week 124 | 1.50 (1.04) | 3.24 (8.32)
  Week 128: number analyzed (Participants) | 2 | 15
  Week 128 | 0.65 (0.64) | 3.09 (7.52)
  Week 132: number analyzed (Participants) | 2 | 15
  Week 132 | 2.55 (1.77) | 2.66 (5.04)
  Week 136: number analyzed (Participants) | 2 | 15
  Week 136 | 2.70 (1.27) | 2.85 (7.29)
  Week 140: number analyzed (Participants) | 1 | 13
  Week 140 | 2.50 (NA) — SD was not calculable for 1 participant. | 4.54 (9.57)
  Week 144: number analyzed (Participants) | 2 | 11
  Week 144 | 2.65 (2.19) | 0.96 (1.75)
  Week 148: number analyzed (Participants) | 2 | 12
  Week 148 | 4.80 (0.99) | 0.87 (1.44)
  Week 152: number analyzed (Participants) | 1 | 12
  Week 152 | 1.20 (NA) — SD was not calculable for 1 participant. | 0.79 (0.79)
  Week 156: number analyzed (Participants) | 1 | 11
  Week 156 | 1.80 (NA) — SD was not calculable for 1 participant. | 0.71 (1.17)
  Week 160: number analyzed (Participants) | 1 | 11
  Week 160 | 1.20 (NA) — SD was not calculable for 1 participant. | 0.82 (1.36)
  Week 164: number analyzed (Participants) | 1 | 11
  Week 164 | 1.30 (NA) — SD was not calculable for 1 participant. | 0.54 (0.50)
  Week 168: number analyzed (Participants) | 1 | 10
  Week 168 | 1.30 (NA) — SD was not calculable for 1 participant. | 0.37 (0.22)
  Week 172: number analyzed (Participants) | 1 | 7
  Week 172 | 1.30 (NA) — SD was not calculable for 1 participant. | 0.19 (0.09)
  Week 176: number analyzed (Participants) | 1 | 7
  Week 176 | 1.30 (NA) — SD was not calculable for 1 participant. | 0.25 (0.17)
  Week 180: number analyzed (Participants) | 1 | 7
  Week 180 | 1.20 (NA) — SD was not calculable for 1 participant. | 0.27 (0.16)
  Week 184: number analyzed (Participants) | 1 | 6
  Week 184 | 1.10 (NA) — SD was not calculable for 1 participant. | 0.22 (0.11)
  Week 188: number analyzed (Participants) | 1 | 4
  Week 188 | 2.40 (NA) — SD was not calculable for 1 participant. | 0.21 (0.13)
  Week 192: number analyzed (Participants) | 1 | 2
  Week 192 | 1.10 (NA) — SD was not calculable for 1 participant. | 0.33 (0.25)
  Week 196: number analyzed (Participants) | 1 | 2
  Week 196 | 2.00 (NA) — SD was not calculable for 1 participant. | 0.15 (0.00)
  Week 200: number analyzed (Participants) | 1 | 1
  Week 200 | 1.10 (NA) — SD was not calculable for 1 participant. | 0.50 (NA) — SD was not calculable for 1 participant.
  Week 204: number analyzed (Participants) | 0 | 1
  Week 204 |  | 0.15 (NA) — SD was not calculable for 1 participant.
  Week 208: number analyzed (Participants) | 1 | 0
  Week 208 | 1.00 (NA) — SD was not calculable for 1 participant. |
  Week 212: number analyzed (Participants) | 1 | 0
  Week 212 | 1.60 (NA) — SD was not calculable for 1 participant. |
  Week 216: number analyzed (Participants) | 1 | 0
  Week 216 | 1.10 (NA) — SD was not calculable for 1 participant. |

32. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies to Satralizumab in the DB Period
Description: Reported here is the percentage of participants with at least one positive anti-drug antibody measurement during the DB period.
Time Frame: Up to approximately Week 216
Population: Participants from SAF who received satralizumab were evaluated for this outcome measure. The SAF included all randomized participants who had received at least 1 dose of satralizumab or placebo. Data was summarized together for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Satralizumab, Then Satralizumab
Number analyzed (Participants) | 63
percentage of participants | 71.4

ADVERSE EVENTS:
Time Frame: Double Blind Period: Up to primary clinical cut-off date, 12 Oct 2018 (up to approximately 217 weeks) Open Label Period: Up to primary clinical cut-off date, 31-Jan-2022 (up to approximately 336 weeks)
Description: The SAF included all randomized participants who had received at least 1 dose of satralizumab or placebo.
Groups:
- Placebo Double Blind Period: Participants received matching placebo, subcutaneous (SC) injection at Weeks 0, 2 and 4, and every 4 weeks (Q4W) thereafter throughout the double-blind (DB) period. Participants who experienced a protocol defined relapse could continue in the Open Label Extension (OLE) period 31 days after relapse. Participants who completed the DB period without relapse could participate in the OLE period 4 weeks after receiving their last dose in the DB period.
- SA237 Double Blind Period: Participants received satralizumab 120 mg subcutaneous (SC) injection at Weeks 0, 2 and 4, and every 4 weeks (Q4W) thereafter throughout the double-blind (DB) period. Participants who experienced a protocol defined relapse could continue in the Open Label Extension (OLE) period 31 days after relapse. Participants who completed the DB period without relapse could participate in the OLE period 4 weeks after receiving their last dose in the DB period.
- Placebo Open Label Period: Participants received matching placebo, subcutaneous (SC) injection at Weeks 0, 2 and 4, and every 4 weeks (Q4W) thereafter throughout the double-blind (DB) period. Following the DB period, all participants received satralizumab 120 mg SC injection at Weeks 0, 2 and 4, and Q4W thereafter up to the clinical cut-off date (CCOD).
- SA237 Open Label Period: Participants received satralizumab 120 mg subcutaneous (SC) injection at Weeks 0, 2 and 4, and every 4 weeks (Q4W) thereafter throughout the double-blind (DB) period. Following the DB period, all participants received satralizumab 120 mg SC injection at Weeks 0, 2 and 4, and Q4W thereafter up to the clinical cut-off date (CCOD).
Arm/Group | Placebo Double Blind Period | SA237 Double Blind Period | Placebo Open Label Period | SA237 Open Label Period
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/63 | 0/28 | 0/56
Serious Adverse Events (participants affected / at risk) | 5/32 | 12/63 | 3/28 | 7/56
Other Adverse Events (participants affected / at risk) | 23/32 | 57/63 | 23/28 | 42/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Double Blind Period (N=32) | SA237 Double Blind Period (N=63) | Placebo Open Label Period (N=28) | SA237 Open Label Period (N=56)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuromyelitis optica pseudo relapse (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Double Blind Period (N=32) | SA237 Double Blind Period (N=63) | Placebo Open Label Period (N=28) | SA237 Open Label Period (N=56)
Neutropenia (Blood and lymphatic system disorders) | 1 (10) | 4 (5) | 2 (3) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 5 (19) | 1 (1) | 3 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (6) | 11 (15) | 1 (1) | 3 (4)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 2 (3)
Cellulitis (Infections and infestations) | 0 (0) | 4 (5) | 0 (0) | 2 (4)
Influenza (Infections and infestations) | 2 (3) | 3 (3) | 4 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 9 (11) | 5 (8) | 6 (8)
Oral candidiasis (Infections and infestations) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (14) | 10 (20) | 8 (19) | 10 (32)
Urinary tract infection (Infections and infestations) | 8 (23) | 11 (36) | 5 (8) | 10 (23)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 4 (4) | 0 (0) | 4 (10)
Alanine aminotransferase increased (Investigations) | 0 (0) | 4 (4) | 1 (2) | 1 (1)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (2) | 3 (5) | 4 (9)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 4 (5) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (4) | 2 (6) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2) | 1 (1) | 1 (6) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 5 (9) | 1 (1) | 3 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 14 (14) | 3 (3) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (5) | 3 (3) | 4 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5) | 1 (1) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 9 (12) | 2 (2) | 7 (11)
Balance disorder (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 3 (3) | 2 (3) | 5 (6)
Headache (Nervous system disorders) | 4 (5) | 10 (13) | 4 (4) | 8 (12)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 5 (6) | 2 (2) | 4 (5)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 6 (10) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 6 (6) | 3 (4) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 3 (3) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 1 (1) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (9) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 10 (16) | 3 (3) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (3) | 1 (1) | 3 (3)
Blood fibrinogen decreased (Investigations) | 0 (0) | 1 (4) | 3 (4) | 4 (5)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Complement factor decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 5 (10)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Low density lipoprotein increased (Investigations) | 1 (1) | 1 (1) | 2 (6) | 2 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (14)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (3) | 7 (9) | 1 (1) | 2 (2)
Influenza like illness (General disorders) | 1 (3) | 2 (5) | 1 (1) | 3 (13)
Injection site erythema (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Complement factor C4 decreased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Prothrombin time prolonged (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT02073279/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/79/NCT02073279/SAP_001.pdf